CLINICAL TRIAL: NCT07257887
Title: Assessment of the Efficacy and Safety of OROXID® Oral Solution in Patients With Periodontitis
Acronym: OroxParodont
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ENIKAM d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OROXID-PR-02-25
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Disease
Keywords: Periodontal Disease; hydrogen peroxide; mouth rinses
MeSH Terms: conditions — Periodontal Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OROXID® forte oral solution (Experimental): Medical device: OROXID® forte oral solution
  Interventions: Device: OROXID® forte oral solution
- OROXID® sensitive oral solution (Experimental): Medical device: OROXID® sensitive oral solution
  Interventions: Device: OROXID® sensitive oral solution
- Standard of Care (Other): Oral solutions are not allowed
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: OROXID® forte oral solution — Patients will use OROXID® forte oral solution two to three times daily for 12 weeks as an adjunct to standard care.
  Arms: OROXID® forte oral solution
Device: OROXID® sensitive oral solution — Patients will use OROXID® sensitive oral solution two to three times daily for 12 weeks as an adjunct to standard care.
  Arms: OROXID® sensitive oral solution
Other: Standard of Care — Patients will receive standard of care, consisting of proper tooth brushing without the use of any mouthwash or other products intended to maintain oral hygiene or reduce oral bacterial load.
  Arms: Standard of Care

SUMMARY:
Periodontitis is a chronic, irreversible inflammatory disease affecting the supporting structures of the teeth. It is most commonly caused by bacteria in dental plaque, also known as biofilm. The disease typically begins as gingivitis, a reversible inflammation of the gums resulting from plaque accumulation. Without appropriate intervention-such as maintaining proper oral hygiene and removing plaque-gingivitis can progress to periodontitis, leading to the loss of clinical attachment, alveolar bone resorption, and eventually tooth loss.

Early diagnosis and regular treatment of periodontal disease are essential to prevent disease progression. The treatment of periodontitis is primarily causal and involves the mechanical removal of plaque. Initial therapy is non-surgical, consisting of scaling and root planing, and may be followed by surgical procedures if required. In addition to mechanical cleaning, increasing attention has been given to adjunctive, non-invasive therapies such as mouth rinses or oral solutions containing chlorhexidine or hydrogen peroxide. These agents have antimicrobial properties, help reduce plaque accumulation, and support tissue healing.

Hydrogen peroxide mouth rinses have been used for more than a century as an adjunct to mechanical plaque removal and for the prevention or management of oral infections. However, despite their long history of use, clinical studies evaluating hydrogen peroxide-based mouth rinses remain limited and heterogeneous in design, which makes it difficult to compare findings across studies.

The objective of this post-marketing clinical study is to generate additional data on the safety and efficacy of a hydrogen peroxide mouth rinse as an adjunctive therapy in the treatment of periodontitis. The study will evaluate two hydrogen peroxide concentrations: a 1.5% solution (Oroxid® sensitive) and a 3% solution (Oroxid® forte).

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy participants aged 18 years or older.
2. Generalized periodontitis, Stage III, Grade B.
3. Presence of three or more periodontal pockets deeper than 5 mm.
4. At least 16 natural teeth (excluding wisdom teeth).
5. Ability to comply with oral hygiene instructions following the intervention.
6. Signed informed consent form after being fully informed about the study.

Exclusion Criteria:

1. Periodontal treatment within the past six months.
2. Dental procedures (surgery, professional cleaning, scaling and root planing, laser therapy, piezotome) within the past six months.
3. Periodontitis, Stage IV.
4. Use of mouth rinses or oral gels within the past month.
5. Use of antibiotic therapy within the past three months.
6. Ongoing therapy with antihypertensives, antilipemics, antiarrhythmics, or other cardiovascular medications.
7. Systemic diseases such as diabetes, HIV/AIDS, liver diseases, chronic kidney disease, tuberculosis, and autoimmune disorders (e.g., lupus, scleroderma, Crohn's disease).
8. History of cardiovascular diseases, including acute myocardial infarction, angina pectoris, heart failure, atrial fibrillation, atrioventricular block, peripheral artery disease, or stroke.
9. Therapy with immunosuppressive agents.
10. Allergy to any ingredients of the study products.
11. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Probing depth | Baseline and Week 12
  Mean change in probing depth (measured in millimeters) from baseline to Week 12, comparing the two active treatment groups (OROXID® forte and OROXID® sensitive) with the control group. Probing Depth is the measurement of the distance from the gingival margin to the bottom of the periodontal pocket using a periodontal probe. Values typically range from 1-3 mm (healthy) to ≥5 mm (indicative of periodontal disease), with deeper pockets reflecting more severe attachment loss.
Bleeding on Probing (BOP) | Baseline and Week 12
  Difference in the presence of bleeding on probing (BOP) between the two active treatment groups and the control group after 12 weeks of treatment. BOP evaluates gingival inflammation by recording the presence/absence of bleeding within 30 seconds after gentle periodontal probing, serving as a key diagnostic indicator of active periodontal disease.

SECONDARY OUTCOMES:
Gingival Index (GI) | Baseline and Week 12
  Mean change in Gingival Index (Silness and Löe) scores from baseline to Week 12, comparing the two active treatment groups (OROXID® forte and OROXID® sensitive) with the control group. The Gingival Index (GI) evaluates the severity of gingival inflammation on a scale of 0 to 3, based on redness, swelling, and bleeding on probing.
Plaque Index (PI) | Baseline and Week 12
  Differences in Plaque Index (PI) scores between the active and control groups will be evaluated using the Silness and Löe Plaque Index. This index assesses the thickness of dental plaque along the gingival margin based on the following scoring criteria: Score 0 = No plaque score; 1 = Mild plaque along the gingival margin; Score 2 =Moderate layer of plaque along gingival margin, interdental spaces free; Score 3 = Abundant plaque along the gingival margin, interdental spaces filled with plaque. Higher scores indicate poorer oral hygiene and greater plaque accumulation.
Rate of infection | Up to week 12
  Incidence of infections in each group
Adverse events | Throughout the 12-week study period
  Number and percentage of participants experiencing adverse events (AEs) related to the use of OROXID® forte or OROXID® sensitive during the 12-week study period. The nature, severity, and relationship of each AE to the study product will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Urban Matoh, DMD, Principal Investigator — Klinika Križaj Ljubljana
Locations (2):
- Slovenia (2):
  - Klinika Križaj Ljubljana, Ljubljana
  - Ustna medicina d.o.o., Ljubljana

IPD SHARING:
Plan to Share IPD: No
As a company operating under the jurisdiction of the EU, the organization is subject to the General Data Protection Regulation (GDPR), which imposes strict requirements on the processing and sharing of personal data, including health-related information. Individual Participant Data (IPD) from clinical trials is considered sensitive personal data under GDPR.
  Even when data is anonymized or pseudonymized, sharing IPD with third parties-especially outside the EU-requires careful assessment of data protection safeguards, appropriate legal basis, and in some cases, additional participant consent. Unless all conditions for lawful data transfer and processing are met, including compliance with GDPR Articles 44-50 concerning international data transfers, the sharing of IPD is not permitted.
  For this reason, and to ensure full compliance with EU data protection regulations while safeguarding the privacy and rights of study participants, individual-level data cannot currently be shared.